CLINICAL TRIAL: NCT01287624
Title: A Phase III, Multicenter, Open-Label, Randomized Study of Gemcitabine Plus Cisplatin (GP) Versus Gemcitabine Plus Paclitaxel (GT) as First-Line Treatment in Patients With Advanced Triple-Negative Breast Cancer
Brief Title: Gemcitabine Plus Cisplatin Versus Gemcitabine Plus Paclitaxel in Triple Negative Breast Cancer (TNBC)
Acronym: TNBC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: 307 Hospital of PLA (Other); The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other); Sun Yat-sen University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Zhejiang Cancer Hospital (Other); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xichun Hu, Dr, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2010-04; CBCSG 006 (Other: Chinese Breast Cancer Study Group)
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: triple negative breast cancer; fine line chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Gemcitabine; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine,cisplatin (Experimental): GP (gemcitabine and cisplatin)
  Interventions: Drug: Gemcitabine,cisplatin
- Gemcitabine, Paclitaxel (Active Comparator): GT (gemcitabine and paclitaxel combination)
  Interventions: Drug: Gemcitabine, Paclitaxel

INTERVENTIONS:
Drug: Gemcitabine,cisplatin — Gemcitabine 1250 mg/m2, IV drip 30 minutes, D1, D8 Cisplatin 75 mg/m2, IV drip 120 minutes, D1
  Other Names: experimental arm
  Arms: Gemcitabine,cisplatin
Drug: Gemcitabine, Paclitaxel — Gemcitabine 1250 mg/m2, IV drip 30 minutes, D1, D8 Paclitaxel 175 mg/m2, IV, 3h,D1
  Other Names: control arm
  Arms: Gemcitabine, Paclitaxel

SUMMARY:
This is a prospective, multi-center, open-labeled, randomized phase III clinical trial comparing overall response rate (ORR), progression free survival (PFS), overall survival (OS) and toxicity obtained with gemcitabine cisplatin combination (GP) versus gemcitabine paclitaxel combination (GT).

DETAILED DESCRIPTION:
The previous phase II study showed that gemcitabine and cisplatin combination (GP) is an effective regimen in triple negative breast cancer (TNBC). The potential therapeutic effects of GP in advanced TNBC deserve further evaluation yet. Eligible patients are randomly assigned to receive either GP or GT regimen to verify the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 and 70 years old
2. Histological proven unresectable recurrent or advanced breast cancer
3. Triple-negative for estrogen receptor (ER), progestogen receptor (PR), and human epithelial receptor-2 (HER2) by immunohistochemistry (IHC) test. For patients with ER negative, PR negative, Her2 two plus, a negative Her2 gene amplification should be verified with FISH test. Her2 one plus may consider FISH verification.
4. No prior chemotherapy for metastatic breast cancer. Prior use of taxanes in the adjuvant/neoadjuvant setting is acceptable if completed 6 months prior to enrollment
5. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST)
6. Performance status not more than 1
7. All patients enrolled are required to have adequate hematologic, hepatic, and renal function
8. Life expectancy greater than 12 weeks
9. No serious medical history of heart, lung, liver and kidney
10. Provision of written informed consent prior to any study specific procedures
11. Patients with good compliance

Exclusion Criteria:

1. Pregnant or lactating women (female patients of child-bearing potential must have a negative serum pregnancy test within 14 days of first day of drug dosing, or, if positive, a pregnancy ruled out by ultrasound)
2. Women of child-bearing potential, unwilling to use adequate contraceptive protection during the course of the study
3. Treatment with radiotherapy at the axial skeleton within 4 weeks before the first treatment or has not recovered from all toxicities of previously administered radiotherapy
4. Treatment with an investigational product within 4 weeks before the first treatment
5. Symptomatic central nervous system metastases, except for patients with stable and asymptomatic brain metastases who have completed a course of cranial irradiation, and have at least one measurable lesion outside the brain. Radiotherapy should be completed within 4 weeks prior to the registration
6. Other active malignancies (including other hematologic malignancies) or other malignancies within the last 5 years, except for cured nonmelanoma skin cancer or cervical intraepithelial neoplasia.
7. Patient having a history of clinically significant cardiovascular, hepatic, respiratory or renal diseases, clinically significant hematological and endocrinal abnormalities, clinically significant neurological or psychiatric conditions
8. Uncontrolled serious infection

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
PFS (Progression Free Survival) | 6 weeks

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang J, Lin Y, Sun XJ, Wang BY, Wang ZH, Luo JF, Wang LP, Zhang S, Cao J, Tao ZH, Wu J, Shao ZM, Yang WT, Hu XC. Biomarker assessment of the CBCSG006 trial: a randomized phase III trial of cisplatin plus gemcitabine compared with paclitaxel plus gemcitabine as first-line therapy for patients with metastatic triple-negative breast cancer. Ann Oncol. 2018 Aug 1;29(8):1741-1747. doi: 10.1093/annonc/mdy209. PMID 29905759
- [Derived] Hu XC, Zhang J, Xu BH, Cai L, Ragaz J, Wang ZH, Wang BY, Teng YE, Tong ZS, Pan YY, Yin YM, Wu CP, Jiang ZF, Wang XJ, Lou GY, Liu DG, Feng JF, Luo JF, Sun K, Gu YJ, Wu J, Shao ZM. Cisplatin plus gemcitabine versus paclitaxel plus gemcitabine as first-line therapy for metastatic triple-negative breast cancer (CBCSG006): a randomised, open-label, multicentre, phase 3 trial. Lancet Oncol. 2015 Apr;16(4):436-46. doi: 10.1016/S1470-2045(15)70064-1. Epub 2015 Mar 18. PMID 25795409